CLINICAL TRIAL: NCT04094727
Title: Targeting Malaria High-risk Populations With Tailored Intervention Packages: A Study to Assess Feasibility and Effectiveness in Northern Namibia
Brief Title: Malaria High-Risk Populations in Namibia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: University of Namibia (Other); Ministry of Health and Social Services, Namibia (Other Government); University of Texas Southwestern Medical Center (Other); University of Notre Dame (Other); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Malaria HRP in Namibia
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Malaria
Keywords: malaria; Namibia
MeSH Terms: conditions — Malaria | interventions — Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Presumptive treatment and enhanced vector control (Experimental): For all eligible HRPs in intervention areas, after obtaining informed consent, presumptive treatment for malaria will be carried out using artemether-lumefantrine (AL) at two time points.
  Enhanced vector control activities will include: (1) a mop up indoor residual spraying (IRS) campaign and (2) distribution of long-lasting insecticide-treated nets (LLINs) and/or vector control packs with topical repellent.
  The intervention arm will also receive the standard of care in Namibia.
  Interventions: Drug: Presumptive treatment with Artemether-lumefantrine (AL); Other: Enhanced vector control
- Standard of care (No Intervention): The control arm will receive the standard of care in Namibia: passive case detection through health facilities and health extension workers, routine indoor residual spraying (IRS), and reactive case detection (RACD) accompanied by reactive IRS.

INTERVENTIONS:
Drug: Presumptive treatment with Artemether-lumefantrine (AL) — All eligible HRPs will be presumptively treated with artemether-lumefantrine (AL) at two timepoints, separated by at least one month. All individuals who have provided informed consent, meet eligibility criteria, are not pregnant or breastfeeding, and who do not have symptoms associated with severe malaria or another severe illness, will be offered an age-appropriate course of AL (age-specific blister packages). AL is currently the first line drug used for uncomplicated malaria in Namibia, and has been used previously in northern Namibia for focal mass drug administration and has no severe adverse effects and is well-tolerated, with high adherence and acceptability in this context. AL requires two daily doses for three consecutive days, for a total of six doses. The first antimalarial dose will be delivered by directly observed therapy (DOT) and subsequent doses will be left with the subject, with instructions to self-administer them.
  Other Names: Coartem
  Arms: Presumptive treatment and enhanced vector control
Other: Enhanced vector control — The mop up indoor residual spraying (IRS) campaign will be targeted to farms and cattle posts/kraals in intervention areas in December 2019 to fill gaps from the routine spray campaign (September to November 2019) and utilize the same insecticides and protocols as the national campaign. The team will spray each unsprayed structure with the recommended solution of dichloro-diphenyl-trichloroethane (DDT) for traditional structures and/or Actellic for modern structures, tarps and tents.
  Alternative vector control interventions, including LLINs (long-lasting insecticide treated bed nets), sprayed tents/tarps and topical repellents will be distributed to eligible HRPs between November and January 2020 during one round.
  Other Names: Indoor residual spraying (IRS); Long-lasting insecticide treated bed nets; Topical repellents
  Arms: Presumptive treatment and enhanced vector control

SUMMARY:
This study aims to determine the effectiveness, cost-effectiveness, acceptability, and feasibility of targeted delivery of a package of malaria interventions for improving effective coverage and reducing Plasmodium falciparum malaria transmission among malaria high-risk populations in Northern Namibia. Previous research identified cattle herders and agricultural workers as populations at higher risk of infection. The investigators hypothesize that targeted delivery of interventions will lead improve coverage in these groups and lead to a reduction in P. falciparum transmission.

DETAILED DESCRIPTION:
This study is the second phase of work in Zambezi and Ohangwena Regions, Namibia, building off a formative phase of work that characterized the risk behaviors migratory patterns, health-seeking behaviors, intervention strategies and social networks of agricultural workers and cattle herders, who are previously identified malaria high-risk populations (HRPs). This phase of the study now aims to determine the effectiveness, cost-effectiveness, acceptability, and feasibility of targeted delivery of a package of malaria interventions for improving effective coverage and reducing Plasmodium falciparum malaria transmission in these regions among these populations.

The study will specifically assess the coverage and impact of interventions delivered at worksites to HRPs, including presumptive treatment administered alongside vector control interventions (indoor residual spraying [IRS], long-lasting insecticidal nets [LLINs], and topical repellents). The effectiveness of these interventions will be compared against areas with no study interventions (standard of care) over the course of implementation (November 2019 - May 2020). Primary outcomes will include the coverage of each intervention at worksites over the study period and PCR-based P. falciparum prevalence measured at endline. Following a baseline cross-sectional survey in November/December 2019, the interventions will consist of 2 rounds of presumptive treatment spaced at least one month apart between January and March, and delivery of vector control interventions at worksites and key access points with support from employers, with the primary evaluation to be conducted through an endline cross-sectional survey in April/May 2020. Secondary outcomes around effectiveness will be assessed through incident case data providing measures of incidence in HRP and non-HRP populations, odds of infection associated with each intervention in cases compared to controls and entomological data collection. In addition, operational and feasibility outcomes will be assessed through qualitative data collection, population size estimation of HRP groups and a global positioning system (GPS) logger study.

ELIGIBILITY:
Inclusion Criteria: HRP study populations (all)

* Study participants include those in the 8 selected health facility catchment areas within Zambezi and Ohangwena Regions.
* Identify primary occupation as a agricultural worker or cattle herder
* Zambezi Region: Have slept or worked outside at a farm or cattle post in the past 7 days or will do over the next 3 weeks (sleeping outside, working outside ploughing or guarding crops/cattle, or sleeping in any type of structure located at a farm or cattle post site)
* Ohangwena Region: Report overnight travel to Angola for grazing cattle during the malaria transmission season (November to May) Be willing and able to provide consent (ie mentally fit)

Inclusion Criteria: Presumptive AL treatment

* In addition to the above, subjects must report travel outside of Namibia within the past 60 days to be eligible to receive AL.

Inclusion Criteria: Enhanced vector control

* In addition to the above, participants must not sleep in a structure sprayed with insecticide to be eligible to receive an LLIN or sprayed tent/tarp.

Inclusion Criteria: Focus group discussions and key informant interviews

* Meet eligibility criteria as a member of an HRP, health facility staff or health extension worker involved in the diagnosis and treatment of HRP populations.
* Individuals must be 18 years and older and willing and able to provide consent to be included in the GPS logger, focus group discussions or key informant interviews

Exclusion Criteria:

* Per national guidelines in Namibia, presumptive treatment with AL will not be given to women who are pregnant in the first trimester, individuals weighing less than 5kg, those with a known AL allergy or suspected severe malaria.
* Individuals under the age of 18 will be excluded from the GPS logger study, focus group discussions and key informant interviews.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 3302 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Effective coverage of AL (presumptive treatment) | 6 months, measured post-intervention only
  This is defined as the proportion of eligible HRPs who report receiving a full course of AL (presumptive treatment) at any time over the study period. The difference in intervention coverage between arms at end-line will be assessed using generalized linear models adjusted for potential confounders and a fixed effect to capture clustering at the health facility level.
Effective coverage of IRS | 6 months, measured pre-and post-intervention
  This is defined as the proportion of eligible HRPs who report sleeping at a worksite in a structure sprayed with insecticide during the past 6 months (IRS), at any time over the study period. The difference in intervention coverage between arms will be assessed using a difference-in-difference approach using generalized linear models adjusted for potential confounders and a fixed effect to capture clustering at the health facility level.
Effective coverage of LLIN | 6 months, measured pre-and post-intervention
  This is defined as the proportion of eligible HRPs who report sleeping under a bednet (LLIN) the last night staying at a worksite, at any time over the study period. The difference in intervention coverage between arms will be assessed using a difference-in-difference approach using generalized linear models adjusted for potential confounders and a fixed effect to capture clustering at the health facility level.
Prevalence of infection measured by polymerase chain reaction (PCR) | 6 months
  Species-specific prevalence of malaria infection will be calculated as the proportion of people testing positive for each species malaria by PCR out of all tested HRPs. The reduction in malaria prevalence will be assessed using a difference-in-difference approach, comparing change (pre- versus post-intervention) in all-species infection between intervention and control groups.

SECONDARY OUTCOMES:
Odds of symptomatic malaria associated with receiving each intervention | 6 months
  The odds of clinical malaria associated with receiving each intervention will be measured by comparing the risk of exposure in cases (RDT-positive) to the risk in controls (RDT-negative) in HRPs within study areas.
Total confirmed outpatient (OPD) malaria case incidence by health facility, stratified by HRP status | 6 months
  The total confirmed outpatient malaria case incidence will be estimated for each of the study health catchment areas and stratified by HRP status. RDTs used for routine malaria diagnosis will be collected and a short questionnaire affixed to the back to allow collection of key indicators to stratify incidence estimates. Denominators will be based on health catchment populations and population size estimates obtained through this study. A reduction in malaria incidence in HRPs and the overall catchment population will be evaluated using a difference-in-difference approach, comparing change (pre- versus post-intervention) between intervention and control groups.
Malaria seroprevalence in HRPs | 6 months
  Malaria exposure in HRPs will be measured as the proportion of people with antimalarial antibodies present in their blood serum. ELISA assays will be used to detect biomarkers of Pf exposure, using collected dried blood spots during baseline and endline cross-sectional surveys. The reduction in malaria exposure will be assessed using a difference-in-difference approach, comparing change (pre- versus post-intervention) between intervention and control groups.
Test positivity rates from RACD | 6 months
  Test positivity rates will be calculated as the proportion of individuals screened during routine RACD who test positive for malaria by RDT and PCR. Rates will be stratified by HRP status and location of event (either within villages or at an HRP worksite).Differences in prevalence measures between HRP and non-HRP populations will be assessed using a χ2 test, as well as logistic regression models to account for potential confounding factors.
Entomological Indicators | 6 months
  Entomological measurements including descriptions of vector occurrence, estimates of human biting rates, measures of indoor and outdoor densities, and insecticide susceptibility status and frequency. Measures will be compared between intervention and control study areas, for each type of intervention.
Intervention acceptability as evaluated by participation rate | 6 months
  The acceptability of a targeted delivery of presumptive treatment and vector control interventions to HRPs will be assessed as the proportion of targeted individuals refusing each intervention, among those eligible for inclusion. Acceptability of IRS will be assessed as the proportion of targeted farms refusing LLIN, among those with at least one sprayable structure missed during the spray campaign.
Intervention acceptability as evaluated by qualitative assessment | 6 months
  Qualitative data collection methods such as focus groups and key informant interviews with HRPs, health extension workers, employers and other health sector staff will be implemented to assess intervention acceptability.
Cost effectiveness | 6 months
  The costs and cost-effectiveness of the intervention package will be assessed as an incremental cost effectiveness ratio (ICER), as well as cost per population and case averted as measured through the difference in infections identified subsequent to the intervention. Program data on costs/expenditure for each intervention will be collected and combined with estimates of program effectiveness to estimate these measures.
Adherence to presumptive treatment intervention as evaluated by pill count | 6 months
  Participant adherence to presumptive treatment will be assessed within a sub-sample of people distributed the drug and measured as the proportion of people who complete all pills in the pill pack after receiving the first dose of AL by DOT. Changes in proportions over time will be quantified between the two distribution rounds.
Self-reported compliance to LLIN and topical repellents. | 6 months
  Self-reported user compliance to LLINs and topical repellents will be assessed through the quantitative baseline and endline cross-sectional surveys, as well as through a use tracking log tracking compliance over a 30-day period (Appendix 16 and 17) in the cohort included in the pill count. LLIN use and condition will be empirically assessed during the endline cross-sectional survey and at 30 days, as well as repellent containers weighed after 30 in the cohort. Qualitative information on use of these interventions will be collected during key informant interviews and focus group discussions.
HRP population size | 6 months
  The population size of target HRPs will be estimated in intervention areas using a combination of multiplier and multiple capture-recapture (CR) methods. In Ohangwena Region, the population is assumed fixed, although accessibility of cattle herders in Namibia may vary throughout the year. In Zambezi Region, the population is estimated at two distinct time periods in order to capture turnover between agricultural seasons.
HRP movement patterns | 6 months
  The proportion of individual's time spent in different locations will be measured from aggregating GPS readings (located within pre-defined space-time windows) which are spatially located within a given type of area (farm, cattle post, grazing location, village etc). Where possible, common locations will be tagged and classified by field workers to distinguish individual farms, fields and other points of interests (such as bars, homes, etc). Aggregated GPS readings (located within pre-defined space-time windows) will be plotted to distinguish individual trips and measure specific characteristics of each trip, including distance of travel and frequency of trips.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Smith, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of Namibia, Multidisciplinary Research Centre, Windhoek, Namibia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with any parties outside of the study team.

REFERENCES:
- [Background] Jacobson JO, Cueto C, Smith JL, Hwang J, Gosling R, Bennett A. Surveillance and response for high-risk populations: what can malaria elimination programmes learn from the experience of HIV? Malar J. 2017 Jan 18;16(1):33. doi: 10.1186/s12936-017-1679-1. PMID 28100237
- [Background] Smith JL, Ghimire P, Rijal KR, Maglior A, Hollis S, Andrade-Pacheco R, Das Thakur G, Adhikari N, Thapa Shrestha U, Banjara MR, Lal BK, Jacobson JO, Bennett A. Designing malaria surveillance strategies for mobile and migrant populations in Nepal: a mixed-methods study. Malar J. 2019 May 3;18(1):158. doi: 10.1186/s12936-019-2791-1. PMID 31053075
- [Background] Smith JL, Auala J, Haindongo E, Uusiku P, Gosling R, Kleinschmidt I, Mumbengegwi D, Sturrock HJ. Malaria risk in young male travellers but local transmission persists: a case-control study in low transmission Namibia. Malar J. 2017 Feb 10;16(1):70. doi: 10.1186/s12936-017-1719-x. PMID 28187770
- [Background] Wu L, van den Hoogen LL, Slater H, Walker PG, Ghani AC, Drakeley CJ, Okell LC. Comparison of diagnostics for the detection of asymptomatic Plasmodium falciparum infections to inform control and elimination strategies. Nature. 2015 Dec 3;528(7580):S86-93. doi: 10.1038/nature16039. PMID 26633770
- [Background] Kern SE, Tiono AB, Makanga M, Gbadoe AD, Premji Z, Gaye O, Sagara I, Ubben D, Cousin M, Oladiran F, Sander O, Ogutu B. Community screening and treatment of asymptomatic carriers of Plasmodium falciparum with artemether-lumefantrine to reduce malaria disease burden: a modelling and simulation analysis. Malar J. 2011 Jul 29;10:210. doi: 10.1186/1475-2875-10-210. PMID 21801345
- [Background] Hsiang M, Ntuku H, Roberts K, Dufour M-s, Whittemore B, Tambo M, et al. The effectiveness of malaria reactive focal mass drug administration (rfMDA) and reactive vector control (RAVC), a cluster-randomised controlled two-by-two factorial design trial from the low-endemic setting of Namibi. 2019. Unpublished.
- [Background] Initiative ME. Planning for targeted malaria interventions in high-risk populations (HRPs) in Northern Namibia: Findings from a rapid formative assessment in Zambezi Region. University of California, San Francisco, 2019.
- [Background] The Global Health Group. Screen and treat strategies for malaria elimination: a review of evidence. 2018.
- [Background] Malaria Elimination Initiative. Planning for targeted malaria interventions in high-risk populations (HRPs) in Northern Namibia: Findings from a rapid formative assessment in Ohangwena Region. University of California, San Francisco, 2019.
- [Background] Naing C, Whittaker MA, Tanner M. Inter-sectoral approaches for the prevention and control of malaria among the mobile and migrant populations: a scoping review. Malar J. 2018 Nov 16;17(1):430. doi: 10.1186/s12936-018-2562-4. PMID 30445959
- [Background] IOM (International Organization for Migration). A global report on population mobility and malaria: moving towards elimination with migration in mind. 2013.
- [Derived] Smith JL, Ntuku H, Rerolle F, Burke AM, Mwema T, Turcios K, Uusiku P, Haikali JK, Lifasi M, Smith-Gueye C, Vajda E, Jacobson JO, Greenhouse B, Gosling R, Bennett A, Mumbengegwi DR. Targeting malaria in high-risk populations in low endemic regions in northern Namibia: a quasi-experimental controlled trial to reduce malaria in seasonal agricultural workers and cattle herders. BMJ Glob Health. 2025 Feb 17;10(2):e015565. doi: 10.1136/bmjgh-2024-015565. PMID 39961693